CLINICAL TRIAL: NCT01102101
Title: Effect of Opioids in Neuropathic Pain in Postherpetic Patients
Acronym: VHPRG-HDRPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: WWTF, Wiener Wissenschafts-, Forschungs- und Technologiefonds (Unknown); Vienna General Hospital (Other)
Responsible Party: Professor Burkhard Gustorff, Vienna Human Pain Research Group, Deparmtent of Anaesthesia, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VHPRG-HighDoseRemiPostHerpetic
Record Dates: First submitted 2010-04-06; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Neuralgia, Postherpetic
Keywords: Remifentanil; Hyperalgesia; Zoster; Postherpetic neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic; Hyperalgesia; Herpes Zoster | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Remifentanil — Remifentanil (Ultiva; Glaxo-Smith-Kline; Vienna, Austria) will be applied intravenously during 60 minutes through a dedicated infusion pump (TCI Alaris PK Syringe Pump, Cardinal Health, Baesweiler, Germany), with a Target Controlled Infusion (following the integrated software algorithm by Minto), reaching the initial 18ng/ml plasma concentration in 180 seconds. This corresponds to approx. 0.7 µg kg-1 min-1.
  Other Names: Remifentanil (Ultiva; Glaxo-Smith-Kline; Vienna, Austria)

SUMMARY:
Postherpetic neuralgia (PHN) is often associated with pain and sensory changes and is the leading type of neuropathic pain in modern clinical pain research. It is characterized by a variety of sensory patterns, which may be categorized into "irritable nociceptor" and "impairment of nociceptor". At date, several lines of evidence lead to the assumption, that mechanical hyperalgesia in PHN is based - at least in part - on central nervous processes of sensitization.

In animal studies the investigators have discovered a previously unrecognized effect of opioids, the reversal of long-term potentiation (LTP) at C-fibre synapses, i.e. an opioid-induced depotentiation. In principle, synaptic depotentiation may be permanent or transient. In our study the clinically used ultra-short acting MOR agonist remifentanil normalized synaptic strength after wash-out of the drug. At present it is not known whether opioid-induced depotentiation can be used to the benefit of pain patients.

The aim is to study the hypothesis, that pain in a group of PHN patients with predominant mechanical hyperalgesia is reversed by intravenous remifentanil at a plasma target concentration of 18ng/ml (corresponding to about 0.75 µg/kg/min) for 60 minutes compared with PHN patients of other sensory types.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from PHN.
* Pain ≥ 4 out of 10 in numeric rating scale (NRS)
* Female and male patients above the age of 18
* Ability to understand/write/read german

Exclusion Criteria:

* Zoster affecting trigeminal-, opticus region
* Any somatic pain which is stronger than the neuropathic pain
* Severe progressive disease
* Acute cardiac decompensation
* Known cardiac valve dysfunction
* Known pulmonary hypertension
* Cardiac conduction disturbance
* Active herpetic lesion
* Opioid therapy
* Asthma bronchial
* Chronic obstructive pulmonary disease >GOLD II
* Severe psychiatric condition
* Abuse of alcoholic beverages, drug abuse
* Negative neuropathic symptoms
* Pregnancy or breast feeding
* Participation in a clinical trial in the 2 weeks preceding the study
* Allergy against any medication used in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Stimulus-response (SR)-function | 7 days

SECONDARY OUTCOMES:
Pinprick | 7 days
  Area of secondary hyperalgesia assessed by pinprick
Area of dynamic allodynia | 7 days
  Brush, Q Tip, Cotton Wool
NRS | 7 days
  Pain according to numeric rating scale (NRS)
Mechanical pain threshold | 7 days
  Mechanical pain threshold measured with v. Frey Filaments
HPPT | 7 days
  Heat pain perception threshold (HPPT) with thermal sensory analyzer (TSA)
HPTT | 7 days
  Heat pain tolerance threshold (HPTT) measured with TSA
Coolness | 7 days
  Coolness perception threshold measured with TSA
Warmth | 7 days
  Warmth perception threshold measured with TSA
LDPI | 7 days
  Laser Doppler Perfusion Imager (LDPI) measuring superficial perfusion of the dermatome

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - General Hospital Vienna, Medical University of Vienna, Vienna, Vienna
  - Wilhelminenspital der Stadt WIen, Vienna, Vienna